CLINICAL TRIAL: NCT05514938
Title: Polypill Strategy for Evidence-Based Management of Patients With Acute Coronary Syndrome Undergoing Percutaneous Coronary Intervention in an Underserved Patient Population
Brief Title: Polypill in Acute Coronary Syndrome
Acronym: POLY-ACS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Ambarish Pandey, ASSISTANT PROFESSOR, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU2022-0604
Record Dates: First submitted 2022-08-22; First posted 2022-08-25 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Acute Coronary Syndrome; Lipid Disorder; Coronary Artery Disease
Keywords: Acute coronary syndrome; Antiplatlet therapy; Statin; Lipids; Drug eluting stent
MeSH Terms: conditions — Acute Coronary Syndrome; Lipid Metabolism Disorders; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Polypill (Experimental): Patients will be randomized to receiving a fixed-dose polypill in addition to other guideline-directed medical therapies prescribed by their physician. Polypill formulations will include rosuvastatin 40 mg, aspirin 81 mg, and prasugrel 10 mg daily or rosuvastatin 40 mg, aspirin 81 mg, and clopidogrel 75 mg.
  Interventions: Drug: Polypill
- Usual Care (individual medications prescribed by primary cardiologist) (Active Comparator): Patients will receive usual post-ACS care and medications prescribed by their provider. All of the individual components will be available at low- or no-cost to participants as individual pill formulations.
  Interventions: Drug: Usual Care (individual medications prescribed by primary cardiologist)

INTERVENTIONS:
Drug: Polypill — Polypill formulation consisting of rosuvastatin, aspirin, and prasugrel or consisting of rosuvastatin, aspirin, and clopidogrel.
  Arms: Polypill
Drug: Usual Care (individual medications prescribed by primary cardiologist) — Typical prescriptions for post-acute coronary syndrome care including statin, aspirin, and prasugrel or clopidogrel.
  Arms: Usual Care (individual medications prescribed by primary cardiologist)

SUMMARY:
Acute coronary syndromes (ACS) represent a major contributor to mortality, morbidity, and healthcare costs. Effective therapies are widely available; however, adherence is low. This contributes to worse patient outcomes and increased risk of morbidity and mortality. The once-daily polypill leverages a population-based strategy that has previously demonstrated efficacy in improving adherence and access to therapy in low-resource settings, making it an innovative approach for improving post-ACS care. This study aims to investigate the utility of a polypill-based strategy for patients with ACS with drug eluting stent (DES) placement. The polypill will consist of a high-intensity statin (rosuvastatin 40 mg daily), aspirin 81 mg daily, and either clopidogrel 75 mg or prasugrel 10 mg daily.

DETAILED DESCRIPTION:
Acute coronary syndromes (ACS) represent a large contributor to patient morbidity and mortality and healthcare costs. Patients with suspected ACS are referred for diagnostic coronary angiography, and if obstructive coronary disease is found, percutaneous coronary intervention (PCI) with a drug-eluding stent (DES) has been proven to reduce mortality and reduce recurrent myocardial infarction. Medical therapy for ACS involves treatment with a statin and dual antiplatelet drug therapy with aspirin and P2Y12 inhibition.

Dual antiplatelet therapy (DAPT) is a vital aspect of post-PCI care and ensures stent patency. Aspirin blocks metabolism of arachidonic acid and production of thromboxane A2 through irreversible inhibition of cyclooxygenase 1. Prasugrel and clopidogrel are irreversible inhibitors of the platelet P2Y12 ADP receptors, while ticagrelor is a reversible inhibitor of the platelet P2Y12 ADP receptor. Current guidelines recommend dual antiplatelet therapy for at least 1 month and ideally up to 1 year for patients treated medically, and at least 1 year for patients treated with DES after hospitalization for ACS.

Additionally, lipid lowering therapy is a cornerstone of post-ACS care. Multiple studies have demonstrated a direct correlation between low-density lipoprotein cholesterol (LDL-C) levels and ASCVD risk. Statins (3-hydroxy-3-methylgultaryl-coenzyme A reductase inhibitors) are first-line therapies used to achieve LDL-C reductions. High-intensity statins, such as atorvastatin 40 mg or 80 mg or rosuvastatin 20 mg or 40 mg, can lower LDL-C by > 50%, and patients with history of ACS have greater benefit from high-intensity statins versus low-intensity statins. Importantly, administration of a high-intensity statin is a Class 1 recommendation from the AHA/ACC Non-ST-Elevation ACS guidelines and the ST-Elevation ACS guidelines.

The combination of prompt diagnosis of ACS, management with coronary angiography with possible DES placement, and medical therapy including DAPT has led to improvements in ACS mortality. However, nonadherence to cardiovascular medications is common. Data from the US Veteran's Affair's hospitals show that nearly 30% of patients did not refill clopidogrel after index hospitalization for ACS. In a study of the PREMIER registry, one in seven patients stopped taking clopidogrel therapy after 1 month, and those who stopped had ninefold elevated risk of death within 1 year. Poor adherence to antiplatelet therapy with either aspirin or P2Y12 inhibitors can lead to in-stent thrombosis, a particularly morbid occurrence characterized by high patient morbidity and mortality. Early stoppage of dual antiplatelet therapy increases risk of stent thrombosis 90-fold.

Nonadherence to statins is also well documented. Roughly 1/3 of ischemic heart disease is related to dyslipidemia, and statins are the mainstay of treatment. However, roughly 25-50% of patients discontinue their statin therapy within the first year after treatment initiation. Lipid reduction is a proven strategy to prevent further cardiovascular events, however, medication nonadherence is a significant barrier.

The polypill is a potential strategy for increasing utilization of proven ACS therapies. The polypill refers to a fixed-dose combination of once-daily medication with proven benefits. The feasibility of a polypill-based strategy has been demonstrated for the primary prevention of cardiovascular events. Among patients with hypertension at a federally qualified community health center, the polypill led to a reduction in systolic blood pressure (-7 mm Hg, 95% CI: -2 to -12; p=0.003) and low-density lipoprotein cholesterol (-11 mg/dl, 95% CI: -5 to -18; p=0.0003). Multi-drug combinations have additionally been employed in the Indian Polycap Study, HOPE-3 trial, UMPIRE trial and most recently in the PolyIran study, which demonstrated high rates of adherence, and low rates of adverse events.13-16 In PolyIran, the largest of these studies, more than 6500 healthy individuals were enrolled and randomized to treatment with a polypill containing low doses of a thiazide diuretic, aspirin, statin, and ACE/ARB versus no pharmacologic intervention for primary prevention of cardiovascular disease. Among those receiving the polypill, a 34% risk reduction in major cardiovascular events was observed compared to standard treatment. In the smaller UMPIRE trial, moreover, adherence among participants receiving a polypill formulation was more than three-fold higher than in those receiving usual care. Few studies have enrolled disadvantaged U.S populations to date and no study to our knowledge has evaluated a polypill strategy for treatment of heart failure, where pill burden and adherence continue to present obstacles to improving care.

No randomized trial has evaluated a polypill strategy for the treatment of ACS. Given the significant pill burden and challenges with adherence, a polypill strategy may have substantial advantages. Thus, we have planned a single-center, open-label, pragmatic pilot study of a polypill-based strategy for the treatment of ACS. The polypill will consist of a high-intensity statin (rosuvastatin 40 mg daily), aspirin 81 mg daily, and clopidogrel 75 mg or prasugrel 10 mg daily. The rationale for the trial is summarized as follows:

* Acute coronary syndromes represent a major contributor to mortality, morbidity, and healthcare costs
* Effective therapies are widely available; however, adherence is low. This contributes to worse patient outcomes and increased risk of morbidity and mortality.
* The once-daily polypill leverages a population-based strategy that has previously demonstrated efficacy in improving adherence and access to therapy in low-resource settings, making it an innovative approach for improving post-ACS care.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted with acute coronary syndrome who undergo percutaneous coronary intervention with drug eluting stent placement.

Exclusion Criteria:

1. Age < 18
2. Estimated glomerular filtration rate < 30 mL/min/1.73 m2 as measured by the simplified MDRD formula
3. Current need for inotropes or with cardiac index < 2.2 L/min/m2
4. Current need for systemic anticoagulation
5. Contraindication to receive any components of the polypill
6. History of allergic reaction or intolerance to aspirin, prasugrel or clopidogrel, or rosuvastatin
7. Comorbidities that might be expected to limit lifespan within the 1-month study period
8. Inability to provide written informed consent
9. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Low Density Lipoprotein - Cholesterol | 1 month
  Follow-up LDL-C at 30-days.
Platelet Reactivity | 1 month
  Follow-up platelet reactivity at 30 days. Platelet reactivity was assessed using impedance aggregometry (Ohms, Ω, lower = better platelet inhibition)

SECONDARY OUTCOMES:
Adherence by self-report | 1 month
  Follow-up adherence by Morisky Medication Adherence Scale - 8
Treatment Satisfaction | 1 month
  Follow-up treatment satisfaction by Treatment Satisfaction Questionnaire for Medicine
Quality of Life | 1 month
  Follow-up quality of life by Seattle Angina Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ambarish Pandey, MD, MSCS, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amsterdam EA, Wenger NK, Brindis RG, Casey DE Jr, Ganiats TG, Holmes DR Jr, Jaffe AS, Jneid H, Kelly RF, Kontos MC, Levine GN, Liebson PR, Mukherjee D, Peterson ED, Sabatine MS, Smalling RW, Zieman SJ. 2014 AHA/ACC Guideline for the Management of Patients with Non-ST-Elevation Acute Coronary Syndromes: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2014 Dec 23;64(24):e139-e228. doi: 10.1016/j.jacc.2014.09.017. Epub 2014 Sep 23. No abstract available. PMID 25260718
- [Background] Levine GN, Bates ER, Bittl JA, Brindis RG, Fihn SD, Fleisher LA, Granger CB, Lange RA, Mack MJ, Mauri L, Mehran R, Mukherjee D, Newby LK, O'Gara PT, Sabatine MS, Smith PK, Smith SC Jr. 2016 ACC/AHA Guideline Focused Update on Duration of Dual Antiplatelet Therapy in Patients With Coronary Artery Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines: An Update of the 2011 ACCF/AHA/SCAI Guideline for Percutaneous Coronary Intervention, 2011 ACCF/AHA Guideline for Coronary Artery Bypass Graft Surgery, 2012 ACC/AHA/ACP/AATS/PCNA/SCAI/STS Guideline for the Diagnosis and Management of Patients With Stable Ischemic Heart Disease, 2013 ACCF/AHA Guideline for the Management of ST-Elevation Myocardial Infarction, 2014 AHA/ACC Guideline for the Management of Patients With Non-ST-Elevation Acute Coronary Syndromes, and 2014 ACC/AHA Guideline on Perioperative Cardiovascular Evaluation and Management of Patients Undergoing Noncardiac Surgery. Circulation. 2016 Sep 6;134(10):e123-55. doi: 10.1161/CIR.0000000000000404. Epub 2016 Mar 29. No abstract available. PMID 27026020
- [Background] Bhatt DL, Topol EJ. Scientific and therapeutic advances in antiplatelet therapy. Nat Rev Drug Discov. 2003 Jan;2(1):15-28. doi: 10.1038/nrd985. PMID 12509756
- [Background] Baigent C, Keech A, Kearney PM, Blackwell L, Buck G, Pollicino C, Kirby A, Sourjina T, Peto R, Collins R, Simes R; Cholesterol Treatment Trialists' (CTT) Collaborators. Efficacy and safety of cholesterol-lowering treatment: prospective meta-analysis of data from 90,056 participants in 14 randomised trials of statins. Lancet. 2005 Oct 8;366(9493):1267-78. doi: 10.1016/S0140-6736(05)67394-1. Epub 2005 Sep 27. PMID 16214597
- [Background] Cannon CP, Braunwald E, McCabe CH, Rader DJ, Rouleau JL, Belder R, Joyal SV, Hill KA, Pfeffer MA, Skene AM; Pravastatin or Atorvastatin Evaluation and Infection Therapy-Thrombolysis in Myocardial Infarction 22 Investigators. Intensive versus moderate lipid lowering with statins after acute coronary syndromes. N Engl J Med. 2004 Apr 8;350(15):1495-504. doi: 10.1056/NEJMoa040583. Epub 2004 Mar 8. PMID 15007110
- [Background] Ho PM, Peterson ED, Wang L, Magid DJ, Fihn SD, Larsen GC, Jesse RA, Rumsfeld JS. Incidence of death and acute myocardial infarction associated with stopping clopidogrel after acute coronary syndrome. JAMA. 2008 Feb 6;299(5):532-9. doi: 10.1001/jama.299.5.532. PMID 18252883
- [Background] Spertus JA, Kettelkamp R, Vance C, Decker C, Jones PG, Rumsfeld JS, Messenger JC, Khanal S, Peterson ED, Bach RG, Krumholz HM, Cohen DJ. Prevalence, predictors, and outcomes of premature discontinuation of thienopyridine therapy after drug-eluting stent placement: results from the PREMIER registry. Circulation. 2006 Jun 20;113(24):2803-9. doi: 10.1161/CIRCULATIONAHA.106.618066. Epub 2006 Jun 12. PMID 16769908
- [Background] Iakovou I, Schmidt T, Bonizzoni E, Ge L, Sangiorgi GM, Stankovic G, Airoldi F, Chieffo A, Montorfano M, Carlino M, Michev I, Corvaja N, Briguori C, Gerckens U, Grube E, Colombo A. Incidence, predictors, and outcome of thrombosis after successful implantation of drug-eluting stents. JAMA. 2005 May 4;293(17):2126-30. doi: 10.1001/jama.293.17.2126. PMID 15870416
- [Background] Lemstra M, Blackburn D. Nonadherence to statin therapy: discontinuation after a single fill. Can J Cardiol. 2012 Sep-Oct;28(5):567-73. doi: 10.1016/j.cjca.2012.03.018. Epub 2012 May 31. PMID 22658124
- [Background] Roshandel G, Khoshnia M, Poustchi H, Hemming K, Kamangar F, Gharavi A, Ostovaneh MR, Nateghi A, Majed M, Navabakhsh B, Merat S, Pourshams A, Nalini M, Malekzadeh F, Sadeghi M, Mohammadifard N, Sarrafzadegan N, Naemi-Tabiei M, Fazel A, Brennan P, Etemadi A, Boffetta P, Thomas N, Marshall T, Cheng KK, Malekzadeh R. Effectiveness of polypill for primary and secondary prevention of cardiovascular diseases (PolyIran): a pragmatic, cluster-randomised trial. Lancet. 2019 Aug 24;394(10199):672-683. doi: 10.1016/S0140-6736(19)31791-X. PMID 31448738
- [Background] Munoz D, Uzoije P, Reynolds C, Miller R, Walkley D, Pappalardo S, Tousey P, Munro H, Gonzales H, Song W, White C, Blot WJ, Wang TJ. Polypill for Cardiovascular Disease Prevention in an Underserved Population. N Engl J Med. 2019 Sep 19;381(12):1114-1123. doi: 10.1056/NEJMoa1815359. PMID 31532959
- [Background] Indian Polycap Study (TIPS); Yusuf S, Pais P, Afzal R, Xavier D, Teo K, Eikelboom J, Sigamani A, Mohan V, Gupta R, Thomas N. Effects of a polypill (Polycap) on risk factors in middle-aged individuals without cardiovascular disease (TIPS): a phase II, double-blind, randomised trial. Lancet. 2009 Apr 18;373(9672):1341-51. doi: 10.1016/S0140-6736(09)60611-5. Epub 2009 Mar 30. PMID 19339045
- [Background] Thom S, Poulter N, Field J, Patel A, Prabhakaran D, Stanton A, Grobbee DE, Bots ML, Reddy KS, Cidambi R, Bompoint S, Billot L, Rodgers A; UMPIRE Collaborative Group. Effects of a fixed-dose combination strategy on adherence and risk factors in patients with or at high risk of CVD: the UMPIRE randomized clinical trial. JAMA. 2013 Sep 4;310(9):918-29. doi: 10.1001/jama.2013.277064. PMID 24002278
- [Background] Yusuf S, Bosch J, Dagenais G, Zhu J, Xavier D, Liu L, Pais P, Lopez-Jaramillo P, Leiter LA, Dans A, Avezum A, Piegas LS, Parkhomenko A, Keltai K, Keltai M, Sliwa K, Peters RJ, Held C, Chazova I, Yusoff K, Lewis BS, Jansky P, Khunti K, Toff WD, Reid CM, Varigos J, Sanchez-Vallejo G, McKelvie R, Pogue J, Jung H, Gao P, Diaz R, Lonn E; HOPE-3 Investigators. Cholesterol Lowering in Intermediate-Risk Persons without Cardiovascular Disease. N Engl J Med. 2016 May 26;374(21):2021-31. doi: 10.1056/NEJMoa1600176. Epub 2016 Apr 2. PMID 27040132